CLINICAL TRIAL: NCT01480141
Title: A Therapeutic Trial of Afatinib in the Neoadjuvant Setting. Molecular Effects of Afatinib: A Window of Opportunity Trial In Early Stage NSCLC
Brief Title: A Window of Opportunity Trial of Afatinib In Early Stage Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left MUSC, no patient enrollments
Sponsor: Medical University of South Carolina (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, George R. Simon, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101596
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Study (Experimental): Single arm trial where all patients will be treated with afatinib until the day of surgery and for a minimum of two weeks. Patients will receive treatment with afatinib 40mg orally daily.
  Interventions: Drug: BIBW 2992 (Afatinib)

INTERVENTIONS:
Drug: BIBW 2992 (Afatinib) — Patients will receive treatment with afatinib 40mg orally daily for a minimum of 2 weeks

SUMMARY:
This study is for patients that have Non-Small Cell Lung Cancer (NSCLC) and he or she will have surgery to remove the tumor. The main purpose of this study is to study how safe and suitable treatment with Afatinib is in participants before surgery to remove the tumor. Another goal of the study is to see if treatment with Afatinib affects the growth and activity of the tumor. Afatinib has not been approved for use by the FDA (Food and Drug Administration) and is experimental.

In some persons, the growth of cancer cells is thought to be stimulated by Epidermal Growth Factor (EGF). This is a protein found in the body which binds to the cell wall to sites called receptors and stimulates cell growth. Some cells have too many receptors and uncontrolled growth and because of this, develop into a cancer tumor. There are several other cancer drugs that bind to these receptors to slow or stop cancer growth such as Gefitinib and erlotinib which are FDA approved and used for the treatment of NSCLC.

The drug Afatinib has been shown to inhibit mutated EGF receptors in clinical trials and may be a candidate for the treatment of NSCLC and a variety of early stage cancers. Participants in this study will take Afatinib by mouth, in pill form, for at least 14 days before having their scheduled surgery to remove their cancer tumor. Participants will be observed for side effects and followed for 30 days after surgery to assess the results after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC, who are deemed to be surgical candidates by standard criteria. Patients with all histologies will be allowed to enroll.

Patients with Stage IA to IIIA disease

* ECOG Performance Status 0-1
* Measurable disease by RECIST 1.1 criteria
* Mediastinoscopy and/or Endoscopic Bronchial Ultrasound (EBUS) and/or Endoscopic Ultrasound (EUS) for complete surgical staging when clinically indicated
* Total bilirubin ≤1.5 mg/dl, SGOT (AST) and SGPT (ALT)≥ 3 x ULN
* Serum creatinine ≤ 1.5 mg/dl
* Serious, active infections must be controlled. Patients may be enrolled while still on antibiotics as long as clinical signs of active infection have resolved.
* A signed informed consent document (ICD)
* Patients 18 years or older
* Able and willing to take oral medications

Exclusion Criteria:

* Known preexisting lung disease.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomization.
* Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g. Crohn's disease, malabsorption or CTC grade ≥2 diarrhea of any etiology.
* Baseline (<1 month before treatment) cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram
* Patients may not be receiving any other investigational agents.
* History of allergic reactions to anilinoquinazolins like gefitinib, erlotinib or BIBW 2992
* Uncontrolled intercurrent illness that would preclude a patient from undergoing surgery
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant (positive pregnancy test) or lactating
* Inability to comply with study and/or follow-up procedures
* Patients who are not surgical candidates or refuse surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Feasibility | 30 days post operative care
  The primary endpoint will demonstrate feasibility of neoadjuvant treatment of BIBW 2992 in patients with early stage (IA to IIIA) NSCLC awaiting surgical resection. Feasibility will be assessed based on the ability to complete the treatment for each patient. For our feasibility endpoint we will declare the treatment "completed" if a patient completes at least 14 days of treatment, had a thoracotomy for the planned surgical resection, and 30 days of post operative care.

SECONDARY OUTCOMES:
Safety and Efficacy | 30 post operative care
  The secondary objective is to determine whether pre-operative BIBW 2992 treatment affects metabolic tumor labeling, as measured by PET-CT scanning. We will measure the absolute and the percentage change in SUV from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: George Simon, MD, Principal Investigator — Medical University of South Carolina Hollings Cancer Center
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] Winton T, Livingston R, Johnson D, Rigas J, Johnston M, Butts C, Cormier Y, Goss G, Inculet R, Vallieres E, Fry W, Bethune D, Ayoub J, Ding K, Seymour L, Graham B, Tsao MS, Gandara D, Kesler K, Demmy T, Shepherd F; National Cancer Institute of Canada Clinical Trials Group; National Cancer Institute of the United States Intergroup JBR.10 Trial Investigators. Vinorelbine plus cisplatin vs. observation in resected non-small-cell lung cancer. N Engl J Med. 2005 Jun 23;352(25):2589-97. doi: 10.1056/NEJMoa043623. PMID 15972865
- [Background] Rusch V, Mendelsohn J, Dmitrovsky E. The epidermal growth factor receptor and its ligands as therapeutic targets in human tumors. Cytokine Growth Factor Rev. 1996 Aug;7(2):133-41. doi: 10.1016/1359-6101(96)00016-0. PMID 8899291
- [Background] Jacobs IJ, Skates S, Davies AP, Woolas RP, Jeyerajah A, Weidemann P, Sibley K, Oram DH. Risk of diagnosis of ovarian cancer after raised serum CA 125 concentration: a prospective cohort study. BMJ. 1996 Nov 30;313(7069):1355-8. doi: 10.1136/bmj.313.7069.1355. PMID 8956699
- [Background] Veale D, Kerr N, Gibson GJ, Kelly PJ, Harris AL. The relationship of quantitative epidermal growth factor receptor expression in non-small cell lung cancer to long term survival. Br J Cancer. 1993 Jul;68(1):162-5. doi: 10.1038/bjc.1993.306. PMID 8391303
- [Background] Sekine I, Takami S, Guang SG, Yokose T, Kodama T, Nishiwaki Y, Kinoshita M, Matsumoto H, Ogura T, Nagai K. Role of epidermal growth factor receptor overexpression, K-ras point mutation and c-myc amplification in the carcinogenesis of non-small cell lung cancer. Oncol Rep. 1998 Mar-Apr;5(2):351-4. PMID 9468555
- [Background] Pfeiffer P, Clausen PP, Andersen K, Rose C. Lack of prognostic significance of epidermal growth factor receptor and the oncoprotein p185HER-2 in patients with systemically untreated non-small-cell lung cancer: an immunohistochemical study on cryosections. Br J Cancer. 1996 Jul;74(1):86-91. doi: 10.1038/bjc.1996.320. PMID 8679464
- [Background] Fontanini G, Vignati S, Bigini D, Mussi A, Lucchi H, Angeletti CA, Pingitore R, Pepe S, Basolo F, Bevilacqua G. Epidermal growth factor receptor (EGFr) expression in non-small cell lung carcinomas correlates with metastatic involvement of hilar and mediastinal lymph nodes in the squamous subtype. Eur J Cancer. 1995;31A(2):178-83. doi: 10.1016/0959-8049(93)00421-m. PMID 7718322
- [Background] Reissmann PT, Koga H, Figlin RA, Holmes EC, Slamon DJ. Amplification and overexpression of the cyclin D1 and epidermal growth factor receptor genes in non-small-cell lung cancer. Lung Cancer Study Group. J Cancer Res Clin Oncol. 1999;125(2):61-70. doi: 10.1007/s004320050243. PMID 10190311
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Cappuzzo F, Ligorio C, Toschi L, Rossi E, Trisolini R, Paioli D, Magrini E, Finocchiaro G, Bartolini S, Cancellieri A, Hirsch FR, Crino L, Varella-Garcia M. EGFR and HER2 gene copy number and response to first-line chemotherapy in patients with advanced non-small cell lung cancer (NSCLC). J Thorac Oncol. 2007 May;2(5):423-9. doi: 10.1097/01.JTO.0000268676.79872.9b. PMID 17473658
- [Background] Hirsch FR, Varella-Garcia M, Cappuzzo F, McCoy J, Bemis L, Xavier AC, Dziadziuszko R, Gumerlock P, Chansky K, West H, Gazdar AF, Crino L, Gandara DR, Franklin WA, Bunn PA Jr. Combination of EGFR gene copy number and protein expression predicts outcome for advanced non-small-cell lung cancer patients treated with gefitinib. Ann Oncol. 2007 Apr;18(4):752-60. doi: 10.1093/annonc/mdm003. Epub 2007 Feb 22. PMID 17317677
- [Background] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Background] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125
- [Background] Pao W, Miller V, Zakowski M, Doherty J, Politi K, Sarkaria I, Singh B, Heelan R, Rusch V, Fulton L, Mardis E, Kupfer D, Wilson R, Kris M, Varmus H. EGF receptor gene mutations are common in lung cancers from "never smokers" and are associated with sensitivity of tumors to gefitinib and erlotinib. Proc Natl Acad Sci U S A. 2004 Sep 7;101(36):13306-11. doi: 10.1073/pnas.0405220101. Epub 2004 Aug 25. PMID 15329413
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Cappuzzo F. Erlotinib in gliomas: should selection be based on EGFR and Akt analyses? J Natl Cancer Inst. 2005 Jun 15;97(12):868-9. doi: 10.1093/jnci/dji169. No abstract available. PMID 15956643
- [Background] Tsao MS, Sakurada A, Cutz JC, Zhu CQ, Kamel-Reid S, Squire J, Lorimer I, Zhang T, Liu N, Daneshmand M, Marrano P, da Cunha Santos G, Lagarde A, Richardson F, Seymour L, Whitehead M, Ding K, Pater J, Shepherd FA. Erlotinib in lung cancer - molecular and clinical predictors of outcome. N Engl J Med. 2005 Jul 14;353(2):133-44. doi: 10.1056/NEJMoa050736. PMID 16014883
- [Background] Rosell R, Moran T, Queralt C, Porta R, Cardenal F, Camps C, Majem M, Lopez-Vivanco G, Isla D, Provencio M, Insa A, Massuti B, Gonzalez-Larriba JL, Paz-Ares L, Bover I, Garcia-Campelo R, Moreno MA, Catot S, Rolfo C, Reguart N, Palmero R, Sanchez JM, Bastus R, Mayo C, Bertran-Alamillo J, Molina MA, Sanchez JJ, Taron M; Spanish Lung Cancer Group. Screening for epidermal growth factor receptor mutations in lung cancer. N Engl J Med. 2009 Sep 3;361(10):958-67. doi: 10.1056/NEJMoa0904554. Epub 2009 Aug 19. PMID 19692684
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Takano T, Fukui T, Ohe Y, Tsuta K, Yamamoto S, Nokihara H, Yamamoto N, Sekine I, Kunitoh H, Furuta K, Tamura T. EGFR mutations predict survival benefit from gefitinib in patients with advanced lung adenocarcinoma: a historical comparison of patients treated before and after gefitinib approval in Japan. J Clin Oncol. 2008 Dec 1;26(34):5589-95. doi: 10.1200/JCO.2008.16.7254. Epub 2008 Sep 15. PMID 18794545
- [Background] Zhu JQ, Zhong WZ, Zhang GC, Li R, Zhang XC, Guo AL, Zhang YF, An SJ, Mok TS, Wu YL. Better survival with EGFR exon 19 than exon 21 mutations in gefitinib-treated non-small cell lung cancer patients is due to differential inhibition of downstream signals. Cancer Lett. 2008 Jul 8;265(2):307-17. doi: 10.1016/j.canlet.2008.02.064. Epub 2008 Apr 14. PMID 18407408
- [Background] Sequist LV, Martins RG, Spigel D, Grunberg SM, Spira A, Janne PA, Joshi VA, McCollum D, Evans TL, Muzikansky A, Kuhlmann GL, Han M, Goldberg JS, Settleman J, Iafrate AJ, Engelman JA, Haber DA, Johnson BE, Lynch TJ. First-line gefitinib in patients with advanced non-small-cell lung cancer harboring somatic EGFR mutations. J Clin Oncol. 2008 May 20;26(15):2442-9. doi: 10.1200/JCO.2007.14.8494. Epub 2008 May 5. PMID 18458038
- [Background] Kobayashi S, Boggon TJ, Dayaram T, Janne PA, Kocher O, Meyerson M, Johnson BE, Eck MJ, Tenen DG, Halmos B. EGFR mutation and resistance of non-small-cell lung cancer to gefitinib. N Engl J Med. 2005 Feb 24;352(8):786-92. doi: 10.1056/NEJMoa044238. PMID 15728811
- [Background] Peinado H, Olmeda D, Cano A. Snail, Zeb and bHLH factors in tumour progression: an alliance against the epithelial phenotype? Nat Rev Cancer. 2007 Jun;7(6):415-28. doi: 10.1038/nrc2131. Epub 2007 May 17. PMID 17508028
- [Background] Sabbah M, Emami S, Redeuilh G, Julien S, Prevost G, Zimber A, Ouelaa R, Bracke M, De Wever O, Gespach C. Molecular signature and therapeutic perspective of the epithelial-to-mesenchymal transitions in epithelial cancers. Drug Resist Updat. 2008 Aug-Oct;11(4-5):123-51. doi: 10.1016/j.drup.2008.07.001. Epub 2008 Aug 20. PMID 18718806
- [Background] Thiery JP, Acloque H, Huang RY, Nieto MA. Epithelial-mesenchymal transitions in development and disease. Cell. 2009 Nov 25;139(5):871-90. doi: 10.1016/j.cell.2009.11.007. PMID 19945376
- [Background] Voulgari A, Pintzas A. Epithelial-mesenchymal transition in cancer metastasis: mechanisms, markers and strategies to overcome drug resistance in the clinic. Biochim Biophys Acta. 2009 Dec;1796(2):75-90. doi: 10.1016/j.bbcan.2009.03.002. Epub 2009 Mar 21. PMID 19306912
- [Background] Yilmaz M, Christofori G. Mechanisms of motility in metastasizing cells. Mol Cancer Res. 2010 May;8(5):629-42. doi: 10.1158/1541-7786.MCR-10-0139. Epub 2010 May 11. PMID 20460404
- [Background] Witta SE, Gemmill RM, Hirsch FR, Coldren CD, Hedman K, Ravdel L, Helfrich B, Dziadziuszko R, Chan DC, Sugita M, Chan Z, Baron A, Franklin W, Drabkin HA, Girard L, Gazdar AF, Minna JD, Bunn PA Jr. Restoring E-cadherin expression increases sensitivity to epidermal growth factor receptor inhibitors in lung cancer cell lines. Cancer Res. 2006 Jan 15;66(2):944-50. doi: 10.1158/0008-5472.CAN-05-1988. PMID 16424029
- [Background] Postigo AA, Dean DC. ZEB, a vertebrate homolog of Drosophila Zfh-1, is a negative regulator of muscle differentiation. EMBO J. 1997 Jul 1;16(13):3935-43. doi: 10.1093/emboj/16.13.3935. PMID 9233803
- [Background] Peinado H, Quintanilla M, Cano A. Transforming growth factor beta-1 induces snail transcription factor in epithelial cell lines: mechanisms for epithelial mesenchymal transitions. J Biol Chem. 2003 Jun 6;278(23):21113-23. doi: 10.1074/jbc.M211304200. Epub 2003 Mar 28. PMID 12665527
- [Background] Yang J, Mani SA, Donaher JL, Ramaswamy S, Itzykson RA, Come C, Savagner P, Gitelman I, Richardson A, Weinberg RA. Twist, a master regulator of morphogenesis, plays an essential role in tumor metastasis. Cell. 2004 Jun 25;117(7):927-39. doi: 10.1016/j.cell.2004.06.006. PMID 15210113
- [Background] Bracken CP, Gregory PA, Kolesnikoff N, Bert AG, Wang J, Shannon MF, Goodall GJ. A double-negative feedback loop between ZEB1-SIP1 and the microRNA-200 family regulates epithelial-mesenchymal transition. Cancer Res. 2008 Oct 1;68(19):7846-54. doi: 10.1158/0008-5472.CAN-08-1942. PMID 18829540
- [Background] Bremnes RM, Veve R, Gabrielson E, Hirsch FR, Baron A, Bemis L, Gemmill RM, Drabkin HA, Franklin WA. High-throughput tissue microarray analysis used to evaluate biology and prognostic significance of the E-cadherin pathway in non-small-cell lung cancer. J Clin Oncol. 2002 May 15;20(10):2417-28. doi: 10.1200/JCO.2002.08.159. PMID 12011119
- [Background] Prudkin L, Liu DD, Ozburn NC, Sun M, Behrens C, Tang X, Brown KC, Bekele BN, Moran C, Wistuba II. Epithelial-to-mesenchymal transition in the development and progression of adenocarcinoma and squamous cell carcinoma of the lung. Mod Pathol. 2009 May;22(5):668-78. doi: 10.1038/modpathol.2009.19. Epub 2009 Mar 6. PMID 19270647
- [Background] Hlubek F, Brabletz T, Budczies J, Pfeiffer S, Jung A, Kirchner T. Heterogeneous expression of Wnt/beta-catenin target genes within colorectal cancer. Int J Cancer. 2007 Nov 1;121(9):1941-1948. doi: 10.1002/ijc.22916. PMID 17631641
- [Background] Song J. EMT or apoptosis: a decision for TGF-beta. Cell Res. 2007 Apr;17(4):289-90. doi: 10.1038/cr.2007.25. No abstract available. PMID 17426696
- [Background] Barr S, Thomson S, Buck E, Russo S, Petti F, Sujka-Kwok I, Eyzaguirre A, Rosenfeld-Franklin M, Gibson NW, Miglarese M, Epstein D, Iwata KK, Haley JD. Bypassing cellular EGF receptor dependence through epithelial-to-mesenchymal-like transitions. Clin Exp Metastasis. 2008;25(6):685-93. doi: 10.1007/s10585-007-9121-7. Epub 2008 Jan 31. PMID 18236164
- [Background] Thomson S, Petti F, Sujka-Kwok I, Epstein D, Haley JD. Kinase switching in mesenchymal-like non-small cell lung cancer lines contributes to EGFR inhibitor resistance through pathway redundancy. Clin Exp Metastasis. 2008;25(8):843-54. doi: 10.1007/s10585-008-9200-4. Epub 2008 Aug 12. PMID 18696232
- [Background] Morgillo F, Woo JK, Kim ES, Hong WK, Lee HY. Heterodimerization of insulin-like growth factor receptor/epidermal growth factor receptor and induction of survivin expression counteract the antitumor action of erlotinib. Cancer Res. 2006 Oct 15;66(20):10100-11. doi: 10.1158/0008-5472.CAN-06-1684. PMID 17047074
- [Background] Gemmill RM, Roche J, Potiron VA, Nasarre P, Mitas M, Coldren CD, Helfrich BA, Garrett-Mayer E, Bunn PA, Drabkin HA. ZEB1-responsive genes in non-small cell lung cancer. Cancer Lett. 2011 Jan 1;300(1):66-78. doi: 10.1016/j.canlet.2010.09.007. Epub 2010 Oct 25. PMID 20980099
- [Background] Ohira T, Gemmill RM, Ferguson K, Kusy S, Roche J, Brambilla E, Zeng C, Baron A, Bemis L, Erickson P, Wilder E, Rustgi A, Kitajewski J, Gabrielson E, Bremnes R, Franklin W, Drabkin HA. WNT7a induces E-cadherin in lung cancer cells. Proc Natl Acad Sci U S A. 2003 Sep 2;100(18):10429-34. doi: 10.1073/pnas.1734137100. Epub 2003 Aug 22. PMID 12937339
- [Background] Takeyama Y, Sato M, Horio M, Hase T, Yoshida K, Yokoyama T, Nakashima H, Hashimoto N, Sekido Y, Gazdar AF, Minna JD, Kondo M, Hasegawa Y. Knockdown of ZEB1, a master epithelial-to-mesenchymal transition (EMT) gene, suppresses anchorage-independent cell growth of lung cancer cells. Cancer Lett. 2010 Oct 28;296(2):216-24. doi: 10.1016/j.canlet.2010.04.008. Epub 2010 May 7. PMID 20452118
- [Background] Haura EB, Sommers E, Song L, Chiappori A, Becker A. A pilot study of preoperative gefitinib for early-stage lung cancer to assess intratumor drug concentration and pathways mediating primary resistance. J Thorac Oncol. 2010 Nov;5(11):1806-14. doi: 10.1097/JTO.0b013e3181f38f70. PMID 20881637
- [Background] Lara-Guerra H, Waddell TK, Salvarrey MA, Joshua AM, Chung CT, Paul N, Boerner S, Sakurada A, Ludkovski O, Ma C, Squire J, Liu G, Shepherd FA, Tsao MS, Leighl NB. Phase II study of preoperative gefitinib in clinical stage I non-small-cell lung cancer. J Clin Oncol. 2009 Dec 20;27(36):6229-36. doi: 10.1200/JCO.2009.22.3370. Epub 2009 Nov 2. PMID 19884551
- [Background] Vandesompele J, De Paepe A, Speleman F. Elimination of primer-dimer artifacts and genomic coamplification using a two-step SYBR green I real-time RT-PCR. Anal Biochem. 2002 Apr 1;303(1):95-8. doi: 10.1006/abio.2001.5564. No abstract available. PMID 11906156
- [Background] Warzecha CC, Sato TK, Nabet B, Hogenesch JB, Carstens RP. ESRP1 and ESRP2 are epithelial cell-type-specific regulators of FGFR2 splicing. Mol Cell. 2009 Mar 13;33(5):591-601. doi: 10.1016/j.molcel.2009.01.025. PMID 19285943
- [Background] Shih YC, Xu Y, Cormier JN, Giordano S, Ridner SH, Buchholz TA, Perkins GH, Elting LS. Incidence, treatment costs, and complications of lymphedema after breast cancer among women of working age: a 2-year follow-up study. J Clin Oncol. 2009 Apr 20;27(12):2007-14. doi: 10.1200/JCO.2008.18.3517. Epub 2009 Mar 16. PMID 19289624
- [Background] Kuo SH, Yang CH, Yu CJ, Hsu C, Cheng AL, Yang PC. Survival of stage IIIB/IV non-small cell lung cancer patients who received chemotherapy but did not participate in clinical trials. Lung Cancer. 2005 May;48(2):275-80. doi: 10.1016/j.lungcan.2004.10.004. Epub 2004 Dec 15. PMID 15829329
- [Background] Albanell J, Gascon P. Small molecules with EGFR-TK inhibitor activity. Curr Drug Targets. 2005 May;6(3):259-74. doi: 10.2174/1389450053765888. PMID 15857287
- [Background] Natale RB, Bodkin D, Govindan R, Sleckman BG, Rizvi NA, Capo A, Germonpre P, Eberhardt WE, Stockman PK, Kennedy SJ, Ranson M. Vandetanib versus gefitinib in patients with advanced non-small-cell lung cancer: results from a two-part, double-blind, randomized phase ii study. J Clin Oncol. 2009 May 20;27(15):2523-9. doi: 10.1200/JCO.2008.18.6015. Epub 2009 Mar 30. PMID 19332730
- [Background] Yin JL, Shackel NA, Zekry A, McGuinness PH, Richards C, Putten KV, McCaughan GW, Eris JM, Bishop GA. Real-time reverse transcriptase-polymerase chain reaction (RT-PCR) for measurement of cytokine and growth factor mRNA expression with fluorogenic probes or SYBR Green I. Immunol Cell Biol. 2001 Jun;79(3):213-21. doi: 10.1046/j.1440-1711.2001.01002.x. PMID 11380673